CLINICAL TRIAL: NCT01229046
Title: Pharmacokinetics and Safety of Ticarcillin-clavulanate in Infants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No enrollment occured. Subjects will be enrolled under a new protocol.
Sponsor: Phillip Brian Smith (Other)
Responsible Party: Sponsor-Investigator, Phillip Brian Smith, Associate Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Pro00026692
Record Dates: First submitted 2010-10-14; First posted 2010-10-27 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Sepsis
Keywords: presumed sepsis
MeSH Terms: conditions — Sepsis | interventions — ticarcillin-clavulanic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ticarcillin-clavulanate (Active Comparator): 5 doses of IV ticarcillin-clavulanate infants < 14 days PNA will receive 75 mg/kg Q12 infants ≥ 14 days PNA will receive 75 mg/kg Q8
  Interventions: Drug: Ticarcillin-clavulanic acid

INTERVENTIONS:
Drug: Ticarcillin-clavulanic acid — 5 doses of IV ticarcillin-clavulanate infants < 14 days PNA will receive 75 mg/kg Q12 infants ≥ 14 days PNA will receive 75 mg/kg Q8

SUMMARY:
This study will evaluate the safety, tolerability and PK of ticarcillin-clavulanate in infants <91 days of age with suspected systemic infection.

DETAILED DESCRIPTION:
4.3 Procedures by Visit

4.3.1 Pre-Study Drug Administration Procedures (Study Day 0)

The following procedures will be completed prior to the administration of study drug:

1. Obtain signed and dated informed consent/HIPAA consent
2. Collect demographic data and medical history
3. Perform a complete physical examination
4. Obtain and record infant weight and medication dosing weight for calculation of appropriate study drug dose if different from actual weight
5. Record the following labs if obtained within 72 hours prior to the start of study drug. Use the laboratory values closest to enrollment if there have been multiple tests.

a. Hematology: hematocrit, hemoglobin, white blood cell count with differential, platelet count b. Serum chemistry: glucose, creatinine, blood urea nitrogen, aspartate transaminases (AST), alanine transaminase (ALT), alkaline phosphatase, total and direct bilirubin, sodium, potassium, chloride, calcium, magnesium, total protein, albumin f. Record results of sterile body fluid cultures (blood, urine, CSF, peritoneal fluid) obtained as standard clinical care in the 72 hours prior to study drug administration. Record urine cultures only if obtained by sterile catheterization or suprapubic aspiration g. Document antimicrobials and vasopressors in the 72 hours prior to study drug administration

4.3.2 Procedures During Study Drug Administration (Day 1 to Day 2/3)

1. Record study drug timing of infusion - this includes start/stop times of infusion and amount given
2. Record AEs (definitely and probably related to study drug) from the time of the first dose of study drug
3. Record SAEs from the time of the first dose of study drug
4. Record all concomitant antimicrobials and vasopressors administered
5. Collect blood for PK analysis (see Appendix 2)
6. Record the following labs if obtained in the 72 hours following the 1st dose of study drug. Use the laboratory values closest to the end of this 72 hours period if there have been multiple tests

a. Hematology: hematocrit, hemoglobin, white blood cell count with differential, platelet count b. Serum chemistry: glucose, creatinine, blood urea nitrogen, aspartate transaminases (AST), alanine transaminase (ALT), alkaline phosphatase, total and direct bilirubin, sodium, potassium, chloride, calcium, magnesium, total protein, albumin. (* A serum creatinine must be recorded within (before or after) 72 hours of the 1st dose of study drug) g. Record the results of cultures from sterile body fluids (blood, urine, CSF, peritoneal fluid, or any other sterile body fluid) as obtained per standard of care. Record urine cultures only if obtained by sterile catheterization or suprapubic aspiration

4.3.3 Procedures following Study Drug Administration (Day 3/4 to Day 9/10)

1. Record AEs (definitely and probably related to study drug) for 72 hours following the last dose of study drug
2. Record SAEs for 7 days following the last dose of study drug

4.4 Protocol Deviations When a deviation from the protocol is deemed necessary for an individual infant, the investigator or other responsible physician must contact study PI immediately, unless a delay would endanger the subject, so that a timely decision can be made as to whether or not the infant should be enrolled or continue in the study. The deviation from the protocol will be authorized only for that particular infant. A description of the departure from the protocol and the reason(s) for it must be recorded on the appropriate CRF. Additionally, sites will adhere to local IRB reporting rules for protocol deviations.

5.0 Safety

5.1 Adverse Events

5.1.1 Definition of Adverse Event An AE is defined as any untoward medical occurrence such as a sign(s), symptom (s), and/or laboratory finding(s) concurrent with the use of a drug in humans. AEs include worsening of any baseline symptoms. The event may/may not necessarily have a causal relationship with the administration of the drug. AEs may be reported by the subject, or detected by the investigator, or other competent observer. The investigator will also evaluate any change in laboratory values. If the investigator determines a laboratory abnormality to be clinically significant, it is considered a laboratory AE; however, if the laboratory value abnormality is consistent with a current diagnosis, it may be documented accordingly.

5.1.2 Reporting period AEs (definitely or probably related to study drug) will be recorded from the time of first dose of study drug until 72 hours following the last dose of study drug. All SAEs will be recorded form the time of the first dose of study drug 7 days after the last dose of study drug. The AE reporting period will not be extended if subjects continue on ticarcillin-clavulanate following the 6 doses of study drug. AEs not or possibly related to study drug will NOT be recorded.

5.1.3 Procedures for assessing, recording and reporting AEs Throughout the duration of the study, the investigator will closely monitor each subject for clinical evidence of drug intolerance and monitor all clinically obtained laboratory values for laboratory evidence of AEs. All SAEs will be reported to study's medical monitor within 24 hours. The description of the AE will include description of event, start date, stop date, intensity, if it was serious, and relationship to the study drug. The investigator must verify this information.

The intensity or severity of AEs will be graded as follows:

* Mild - awareness of sign or symptom, but easily tolerated. Not expected to have a clinically significant effect on the subject's overall health and well-being. Not likely to require medical attention
* Moderate - discomfort enough to cause interference with usual activity or affects clinical status. May require medical intervention
* Severe - incapacitating or significantly affecting clinical status. Likely requires medical intervention and/or close follow-up

AEs that increase in intensity will be recorded with a stop date on the AE CRF of the milder AE equal to the date that the condition worsened. A new AE with a start date equal to the date of worsening will then be reported. AEs that decrease in severity need not be reported in this way. The start date will be the date entered above and the date of resolution should be reported as the stop date.

The Investigator is responsible for assessing relationship to study medication using the following definitions:

* Not related: An AE that is due to a pre-existing illness or use of another drug, and is not related to the study drug.
* Possibly related: An AE that has little or no relationship to the study drug and there exists a more likely alternative cause.
* Probably related: An AE that is likely to be related to the administration of the study drug and an alternative cause less likely when compared to the study drug.
* Definitely Related: An AE that has a strong temporal relationship to the study drug. AE will recur with continued or repeated use of the study drug, and another cause is unlikely or less likely.

5.1.4 Follow-up of AEs AEs will be followed until resolution or until stability is reached using good clinical practices.

5.2 Serious Adverse Event

A SAE is defined (21 Code of Federal Regulations part 312.32) as those AEs, which meet any of the following serious outcome criteria:

* Is fatal
* Is life-threatening, meaning, the subject was, in the view of the investigator, at immediate risk of death from the reaction as it occurred, i.e., it does not include a reaction that, had it occurred in a more serious form, might have caused death;
* Is a persistent or significant disability/incapacity, i.e., the event causes a substantial disruption of a person's ability to conduct normal life functions;
* Requires or prolongs inpatient hospitalization;
* Is a congenital anomaly/birth defect;
* Is an important medical event, based on appropriate medical judgment, that may jeopardize the subject or subject may require medical or surgical intervention to prevent one of the other outcomes above.

5.2.1 Procedures for assessing, recording and reporting SAEs All SAEs must be reported by facsimile or electronic transmission to the study's medical monitor within 24 hours after the onset of the SAE (or the awareness of the investigator of the event). The study's medical monitor then notifies the study PI of the SAE within one working day after receiving the report from a clinical site. In addition, a clinical site must report a death or life-threatening event by telephone as soon as possible and within 24 hours to the study's medical monitor.

An SAE CRF must be completed and signed by the site investigator. All SAEs must also be entered into the AE CRF (select "serious").

The FDA requires that all SAEs that are unexpected and potentially related to the study medication must be reported to the FDA in writing within 15 calendar days. SAEs that are unexpected and related to study drug that meet the criteria for death or immediately life-threatening also require the study's medical monitor to notify the FDA by telephone, facsimile transmission or in writing as soon as possible but no later than 7 calendar days, with a follow-up written report within 15 calendar days. The study's medical monitor will prepare an expedited report for the FDA and copies will be distributed to all site investigators. Expedited reports will be placed in the Study Binder by the investigator upon receipt. The investigators will also forward a copy of all expedited reports to their local Investigational Review Boards in accordance with local guidelines.

5.2.2 Follow-up of SAEs All SAEs will be followed until resolution, stabilization or 7 days after the last dose of study drug, whichever occurs, first.

5.3 Blood Volume for PK and Safety Laboratory Tests

Blood sample volume will be minimized by:

1. Most of the hematology and chemistry laboratory measures will be recorded from laboratories drawn as standard of care. Any labs needed for the protocol will count against the total blood volume for the study.
2. A limited PK sampling scheme will be employed such that no more than 1.4 mL of blood (7 samples) is obtained from each subject for PK analysis.

6.0 Administration

6.1 Trial Termination A data safety group with members that have expertise in biostatistics, neonatology, clinical pharmacology, and pediatric infectious disease will monitor the data during the study for AEs, patient safety, and potential toxicity. If two subjects develop an unexpected SAE related to study drug, we will stop enrollment to evaluate the data and safety of the product in this population. Dr. Brian Smith (neonatologist) will receive SAEs and call ad hoc meetings of the safety group as needed.

6.2 Investigational Product

6.2.1 Description of Investigational Product Ticarcillin-clavulanate is a sterile injectable antibacterial combination consisting of the semisynthetic antibiotic ticarcillin disodium, and the β-lactamase inhibitor clavulanate potassium (the potassium salt of clavulanic acid) for intravenous administration. Ticarcillin is derived from the basic penicillin nucleus, 6-amino-penicillanic acid. Clavulanic acid is produced by the fermentation of Streptomyces clavuligerus. It is a β-lactam structurally related to the penicillins and possesses the ability to inactivate a wide variety of β-lactamases by blocking the active sites of these enzymes.

6.3 Drug Accountability Study drug will be provided by the local site pharmacy.

ELIGIBILITY:
Inclusion Criteria:

1. Written permission from parent or legal guardian
2. < 91 days of age
3. < 30 weeks gestation at birth
4. Likely to survive beyond the first 48 hours after enrollment
5. Sufficient intravascular access (either peripheral or central) to receive study drug.

AND ONE OF THE FOLLOWING

* Suspected systemic infection
* Receiving ticarcillin-clavulanate as part of standard of care

Exclusion Criteria:

1. History of allergic reactions to any penicillin, cephalosporins, or beta-lactamase inhibitors
2. Urine output < 0.5 mL/hr/kg over the prior 24 hours
3. Serum creatinine > 1.7 mg/dL
4. Any condition which would make the subject, in the opinion of the investigator, unsuitable for the study

Max Age: 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-09

PRIMARY OUTCOMES:
Clearance of ticarcillin-clavulanate | steady state samples will be drawn on day 2-3 of study drug therapy (around dose 4, 5, or 6)
  The following PK parameters will be estimated:
  1. Systemic clearance
  2. Volume of distribution
  3. Cmax, Tmax, AUC0-Τ, (at steady state), Ke and t1/2
  4. CSF/plasma ticarcillin-clavulanate concentration ratio
  5. Urine/plasma ticarcillin-clavulanate concentration ratio

SECONDARY OUTCOMES:
Incidence of adverse events as a measure of safety and tolerability | 1st dose to 7 days after the last dose
  all serious adverse events and adverse events (definitely and probably related to study drug) will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States